CLINICAL TRIAL: NCT05491005
Title: eHealth Diabetes Remission Trial (Swedish: Remission av Typ 2 Diabetes Med hjälp av eHälsa
Brief Title: The eHealth Diabetes Remission Trial
Acronym: eDIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government); Edgar Sjölunds Diabetes Foundation (Unknown)
Responsible Party: Principal Investigator, Julia Otten, Principal investigator, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2022-02242-01
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Remission; Nutrition Therapy; Obesity; eHealth; Weight Loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Loss | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eHealth (Experimental)
  Interventions: Behavioral: Total diet replacement; Behavioral: eHealth
- Face-to-face (Experimental)
  Interventions: Behavioral: Total diet replacement; Behavioral: Face-to-face
- Healthy control group (No Intervention)

INTERVENTIONS:
Behavioral: Total diet replacement — Total diet replacement (850 kcal/day) for 3 months followed by weight maintenance for 21 months.
  Arms: Face-to-face; eHealth
Behavioral: eHealth — All follow-up through an eHealth application and video meetings.
  Arms: eHealth
Behavioral: Face-to-face — All follow-up through face-to-face meetings.
  Arms: Face-to-face

SUMMARY:
Overweight patients with type 2 diabetes are offered a total diet replacement with the goal of weight loss and diabetes remission. Study participants are randomised to eHealth follow-up or face-to-face follow-up, but the dietary advice is the same in both groups. A healthy control group with normal glucose tolerance is examined once but is not randomised and does not receive any intervention.

DETAILED DESCRIPTION:
One hundred and six overweight patients with type 2 diabetes replace usual foods with total diet replacement (850 kcal/day) for 3 months with the goal of 15 kg weight loss and diabetes remission (HbA1c < 48 mmol/mol without diabetes medication). After 3 months of total diet replacement, food is reintroduced stepwise, and an individually tailored energy prescription is used to prevent weight regain. If study participants do not reach the weight loss goal at 3 months, they are recommended two additional months of total diet replacement. If weight regain occurs during the weight maintenance phase, a rescue plan with total diet replacement will be recommended. To increase the chances to maintain their lower body weight, participants will use a program specifically design for that purpose based on cognitive behavioural therapy. Total study duration is two years.

The one hundred and six participants are randomised to either the eHealth follow-up or the face-to-face follow-up. The dietary advice to achieve and maintain weight loss is the same in both groups and delivered by the same dietician, physician, and nurse but the method of follow-up differs between groups (eHealth vs face-to-face).

eHealth group:

All study information and the cognitive behavioural therapy program is given by an eHealth application in Stöd och behandling which is part of 1177.se. Participants register body weight, fasting blood glucose, and blood pressure every morning at 1177.se. Regularly a measurement of HbA1c is taken at home. Participants will have scheduled video appointments with the study dietician, study nurse or study physician.

Face-to-face group:

Participants have appointments in the medical office with the study physician/nurse/dietician. At the appointments, body weight, blood pressure and capillary blood glucose is measured. HbA1c is measured during the appointments at 0, 6, 12 and 24 months. The cognitive behavioral therapy program for the control group is identical to the program of the intervention group, but the program is delivered during the face-to-face appointments.

Healthy control group:

Fifteen healthy participants with normal glucose tolerance, stable body weight for at least one year and matched to the study participants for sex, age, and weight after one year study duration, will be examined once. These participants are not randomised and do not receive any intervention.

Outcomes:

Primary and secondary outcome measures are compared between 1) the experimental eHealth group and 2) the experimental face-to-face group. For the other pre-specified outcome measures the experimental eHealth group and the experimental face-to-face group are taken together as one group, examined twice (baseline and 12 months) and compared to the healthy control group, that is examined only once.

Long-term follow-up:

Because long term data on diabetes remission by total diet replacement are lacking, study participants will be followed after they have finished the study. Data of the national diabetes registry from participants of this study will be compared to other patients in the national diabetes registry not participating in this study but matched for age, sex and diabetes duration to the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with duration 0-6 years
* BMI 27 kg/m2 and higher
* HbA1c 43 mmol/mol or higher (48 or higher if without diabetes medication)

Exclusion Criteria:

* Insulin treatment
* Weight loss more than 5 kg during the past 6 months
* Diagnosed eating disorder
* eGFR < 30 ml/min/1,73m2
* Myocardial infarction last six months
* Severe heart failure (NYHA class III)
* Ongoing cancer
* Pregnancy
* Treatment with antipsychotic drugs

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 months
  HbA1c without diabetes medication as a continuous outcome (HbA1c correction according to Tsapas et al 2020 if on diabetes medication). The outcome will be tested for non-inferiority first, with a non-inferiority margin of 8 mmol/mol; followed by a test for superiority.

SECONDARY OUTCOMES:
HbA1c | 6 and 24 months
  HbA1c without diabetes medication as a continuous outcome (HbA1c correction according to Tsapas et al 2020 if on diabetes medication). The outcome will be tested for non-inferiority first, with a non-inferiority margin of 8 mmol/mol; followed by a test for superiority.
Diabetes remission | 6, 12 and 24 months
  Number of participants with HbA1c < 48 mmol/mol without diabetes medication. The outcome will be tested for non-inferiority first with a non-inferiority margin of 10 percentage points; followed by a test for superiority.
Body weight | 6, 12 and 24 months
  Body weight as a continuous outcome
Achieved weight loss of at least 15 kg | 6, 12 and 24 months
  Number of participants with achieved weight loss of at least 15 kg
Incremental costs per diabetes remission | 24 months
Estimated lifetime costs | 24 months
Estimated lifetime costs per quality-adjusted life-year (QALY) | 24 months
Fasting blood glucose | 6, 12, 24 months
  Partial diabetes remission (<7.0 mol/l), complete diabetes remission (<6.1 mol/l) without diabetes medication.
P-glucose 120 minutes after the oral glucose tolerance test | 6, 12, 24 months
Number of prescribed oral anti diabetic medications | 6, 12, 24 months
Number of prescribed antihypertensive medications | 6, 12, 24 months
Blood pressure (systolic/diastolic) | 6, 12, 24 months
  Measured at the research facilities
Blood pressure | 6, 12, 24 months
  24h monitoring
Plasma lipid profile | 6, 12, 24 months
Liver enzymes | 6, 12, 24 months
  AST, ALT
Number of participants that discontinue the intervention | 6, 12, 24 months
Waist circumference | 6, 12, 24 months
Relation to food | 6, 12, 24 months
  Three factor eating questionnaire
Estimation of exhaustion | 6, 12, 24 months
  Karolinska Exhaustion Disorder Scale. Minimum value 0. Maximum value 54. A higher score means a worse outcome.
Quality of life accoring to Brunnsviken Brief Quality of Life Scale | 6, 12, 24 months
  The scale estimates how satisfied the participants is with different areas of life, as well as how important each area of life is. Minimum scale 0. Maximum scale 48. A higher score means a better outcome.
Quality of life according to EQ-5D-5L | 6, 12, 24 months
  The questionnaire investigates the dimensions mobility, self-care, usual activities, pain and anxiety/depression. Minimum value 1. Maximum value 5. A higher score means a worse outcome. In addition, a general health score is assessed. Minimum value 0. Maximum value 100. A higher score means a better outcome. All dimension will be analysed separately, but EQ-5D-5L will also be combined to one score.
Eating habits | 6, 12, 24 months
  FFQ 2020 questionnaire
Estimation of health | 6, 12, 24 months
  SF-36 questionnaire
Daily steps | 6, 12, 24 months
  Measured with activity tracker
Study experience | 24 months
  Qualitative questions with written answers about study experience
HbA1c follow-up | Yearly up to 20 years
  Collected from patient journals after study completion
Body weight follow-up | Yearly up to 20 years
  Collected from patient journals after study completion
Blood pressure follow-up | Yearly up to 20 years
  Collected from patient journals after study completion
Usage of diabetes medication follow-up | Yearly up to 20 years
  Collected from patient journals after study completion
Usage of hypertension medication follow-up | Yearly up to 20 years
  Collected from patient journals after study completion
Diabetes complications follow-up | Yearly up to 20 years
  Collected from patient journals and registries after study completion

OTHER OUTCOMES:
Insulin sensitivity | 12 months
  Hyperinsulinemic euglycemic clamp
Insulin secretion | 12 months
  Stepped insulin secretion test with arginine
Metabolic flexibility | 12 months
  Hyperinsulinemic euglycemic clamp
Resting metabolic rate | 12 months
  Indirect calorimetry
Body composition | 12 months
  Dual-energy X-ray absorptiometry (DXA).
Glucagon sensitivity | 12 months
  Plasma amino acids are measured during 120 minutes after a intravenous glucagon bolus
Amino acid tolerance | 12 months
  Plasma amino acids are measured during intravenous amino acid infusion
Glucagon secretion capacity | 12 months
  Plasma glucagon is measured during intravenous amino acid infusion
Gut hormones after carbohydrate intake | 6, 12, 24 months
  GLP-1, GIP and gherkin during the oral glucose tolerance test
P-metabolites and P-lipids after carbohydrate intake | 6, 12, 24 months
  Metabolomics and lipidomics analyses during the oral glucose tolerance test
Liver fat | 12 months
  Measured with MRI
Pancreas fat | 12 months
  Measured with MRI
Fat cell size in subcutaneous fat | 12 months
RNA levels in subcutaneous fat | 12 months
  RNA sequencing
Secretion of adipokines, metabolites and lipids in subcutaneous fat cells ex vivo | 12 months
Plasma testosterone levels | 6, 12 and 24 months
  Only men
Erectile function | 6, 12, 24 months
  Only men, Erectile function subscale
Prostate symptoms | 6, 12, 24 months
  Only men, International prostate symptom score
Urine albumin to creatinine ratio | 6, 12, 24 months
Slow vital capacity (SVC) | 12 months
  Spirometry
Forced vital capacity (FVC) | 12 months
  Spirometry
Forced expiratory volume in 1 s (FEV1) | 12 months
  Spirometry
Diffusion capacity of the the (DCLO) | 12 months
  Spirometry
Experiences of the study participants | Once between 12 and 24 months
  Individual semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Julia Otten, PhD, Principal Investigator — Umeå University
Locations (3):
- Sweden (3):
  - Bra Liv Råslätt vårdcentral, Jönköping
  - Örnsköldsvik hospital, Örnsköldsvik
  - Department of Public Health and Clinical Medicine, Medicine, Umeå

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researchers on reasonable request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data is available to other researchers as soon as it is published.
Access Criteria: Data will be shared with other researchers on reasonable request.

REFERENCES:
- [Background] Tsapas A, Avgerinos I, Karagiannis T, Malandris K, Manolopoulos A, Andreadis P, Liakos A, Matthews DR, Bekiari E. Comparative Effectiveness of Glucose-Lowering Drugs for Type 2 Diabetes: A Systematic Review and Network Meta-analysis. Ann Intern Med. 2020 Aug 18;173(4):278-286. doi: 10.7326/M20-0864. Epub 2020 Jun 30. PMID 32598218
- [Derived] Otten J, Tellstrom A, Schien C, Chninou Y, Lindholm L, Winkvist A, Liv P, Stomby A. eHealth versus face-to-face support for remission of type 2 diabetes by calorie restriction (eHealth DIabetes remission Trial): study protocol for a non-inferiority parallel group randomised controlled trial. BMJ Open. 2025 Jul 22;15(7):e095100. doi: 10.1136/bmjopen-2024-095100. PMID 40701606